CLINICAL TRIAL: NCT04667468
Title: Cold Stored Platelet Early Intervention in Hemorrhagic Shock (CriSP-HS) Trial
Brief Title: Cold Stored Platelet in Hemorrhagic Shock
Acronym: CriSP-HS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21100002; W81XWH-16-D-0024 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-11-24; First posted 2020-12-14 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Trauma; Hemorrhage
Keywords: platelet; hemorrhagic shock; trauma
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Shock, Hemorrhagic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: permuted block design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cold-stored Platelet (CSP) (Experimental): early infusion of one apheresis unit urgent release cold stored platelets (CSP)
  Interventions: Biological: Cold Stored Platelets (CSP)
- Standard Care (Active Comparator): resuscitation, blood and blood component transfusion per site standard care
  Interventions: Biological: Standard Care

INTERVENTIONS:
Biological: Cold Stored Platelets (CSP) — early infusion of urgent release CSP
  Arms: Cold-stored Platelet (CSP)
Biological: Standard Care — standard care including blood and blood component therapy
  Arms: Standard Care

SUMMARY:
The Cold Stored Platelet Early Intervention in Hemorrhagic Shock (CriSP-HS) trial is a proposed 3 year, open label, multi-center, randomized trial designed to determine the feasibility, efficacy, and safety of urgent release cold stored platelets (CSP) in patients in hemorrhagic shock. Patients will be randomized to receive either standard care or early infusion of urgent release cold stored platelets (CSP). The proposed pilot study will utilize 5 level-1 trauma centers from within the LITES network and will enroll approximately 200 patients. The primary outcome for the pilot trial is feasibility, with principal secondary clinical outcome of 24 hour mortality.

DETAILED DESCRIPTION:
The acute management of the severely injured patient with hemorrhage following trauma center arrival has evolved over the last decade.

Current treatment priorities include prevention of coagulopathy through minimization of crystalloid and early blood component resuscitation including plasma and platelets in equal ratios with packed red blood cells. These in-hospital practices, termed damage control resuscitation, are widely used in both battlefield and civilian resuscitation following traumatic injury.

Initiation of the tenets of damage control resuscitation early, soon after arrival, has the potential to reduce downstream complications attributable to hemorrhage by intervening closer to the time of injury, prior to the development of coagulopathy; irreversible shock; and the ensuing inflammatory response. Other blood constituents have recently been shown to be beneficial when given early. Thawed plasma transfusion has been shown to safely reduce 30-day mortality when infused early, in the prehospital setting, in patients at risk of hemorrhagic shock and this separation of survival occurs within the first 3 hours. Platelet transfusion is associated with improved outcomes in the acutely bleeding patients. Cold Stored Platelets have been reported to reduce blood loss when provided for hemorrhage and are a more effective hemostatic product.

Cold stored platelets are less likely to become bacterial contaminated and were the standard of care platelet product until the 1980s. Despite this history and potential benefits, the risks associated with urgent release cold stored platelets and their respective efficacy and function over time are not known in patients with hemorrhagic shock.

By providing Cold Stored Platelets in an urgent release fashion following injury, a potentially superior hemostatic agent is given early, closer to the time of injury. The current pilot trial was designed to determine the feasibility, efficacy and safety of urgent release cold stored platelets as compared to standard care in injured patients in hemorrhagic shock. There are no high-level data which appropriately characterize the urgent release use of cold stored platelets out to 14 days or their function over that time period as compared to standard room temperature platelets. These results will be able to inform future large randomized clinical trials allowing the most appropriate injured population, inclusion criteria, and primary outcome to be selected and utilized.

ELIGIBILITY:
Inclusion Criteria:

Patients with traumatic injury who meet the following criteria:

1. Has 2 or more of any of the following:

   1. Hypotension (systolic blood pressure ≤ 90 mmHg) in the prehospital or emergency department setting
   2. Penetrating mechanism
   3. Abdominal or Extended Focused Assessment with Sonography for Trauma (FAST) abdominal ultrasound is positive or equivocal or deferred by clinical team due to emergent visit to Interventional Radiology or a need for emergent laparotomy, thoracotomy, or vascular exploration
   4. Heart rate ≥ 120 in the prehospital or emergency department setting

   AND
2. Clinical team deems Operating Room (laparotomy, thoracotomy or vascular exploration) or Interventional Radiology for embolization within 60 minutes of arrival to be clinically indicated.

Exclusion Criteria:

1. Wearing "NO CriSP" opt-out bracelet
2. Age >90 or <15 years of age
3. Isolated fall from standing injury mechanism
4. Prisoner
5. Pregnant
6. Traumatic arrest with >5 minutes of CPR without return of vital signs
7. Brain matter exposed or penetrating brain injury (gun shot wound [GSW])
8. Isolated drowning or hanging victims
9. Isolated burns > estimated 20% total body surface area
10. Objection to study voiced by subject or family member in Emergency Department

Inclusion and exclusion criteria will be assessed based on information available at the time of enrollment. If, after subsequent review, it is determined that the subject did not meet inclusion criteria and/or met exclusion criteria, the subject will remain enrolled in the study based on the intent-to-treat principle.

If a verbal report must be used in lieu of physical documentation or directly witnessing inclusion criteria, documentation of the verbal report will serve as the source documentation for determining eligibility.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, MPH, Principal Investigator — University of Pittsburgh; Frank Guyette, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Mississippi, Jackson, Mississippi
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Sciences Center Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the funding agency as well as other researchers upon request to the Principal Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the primary manuscript.
Access Criteria: Requests for data will be submitted in writing and reviewed by the Principal Investigator.

REFERENCES:
- [Derived] Sperry JL, Guyette FX, Rosario-Rivera BL, Kutcher ME, Kornblith LZ, Cotton BA, Wilson CT, Inaba K, Zadorozny EV, Vincent LE, Harner AM, Love ET, Doherty JE, Cuschieri J, Kornblith AE, Fox EE, Bai Y, Hoffman MK, Seger CP, Hudgins J, Mallett-Smith S, Neal MD, Leeper CM, Spinella PC, Yazer MH, Wisniewski SR; Cold Stored Platelet for Hemorrhagic Shock (CRISP-HS) Study Group. Early Cold Stored Platelet Transfusion Following Severe Injury: A Randomized Clinical Trial. Ann Surg. 2024 Aug 1;280(2):212-221. doi: 10.1097/SLA.0000000000006317. Epub 2024 May 6. PMID 38708880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Started | 102 | 98
Completed | 102 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold-stored Platelet (CSP) | Standard Care | Total
Number analyzed (Participants) | 102 | 98 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (14.4) | 34.4 (13.5) | 34.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 85 | 78 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Patients can be in more than one group.
  Participants
    Caucasian | 28 | 18 | 46
    Black | 47 | 51 | 98
    Hispanic | 20 | 13 | 33
    Other including Asian and unknown | 13 | 13 | 26
    Missing | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility
Description: Proportion of eligible patients that can be randomized, enrolled, adhere to protocol, and completed follow-up
Time Frame: Enrollment through 30 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 102 | 98
Participants | 91 | 82

2. Secondary Outcome: 24-hour Mortality
Description: Mortality within 24 hours
Time Frame: Enrollment through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 102 | 98
Participants | 6 | 10

3. Secondary Outcome: 3-hour Mortality
Description: Mortality within 3 hours
Time Frame: Enrollment through 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 102 | 98
Participants | 6 | 7

4. Secondary Outcome: In Hospital Mortality
Description: mortality in-hospital
Time Frame: Enrollment through 30 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 91 | 82
Participants | 12 | 13

5. Secondary Outcome: Hemorrhagic Death Alone
Description: mortality due to hemorrhage
Time Frame: Enrollment through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 102 | 98
Participants | 6 | 7

6. Secondary Outcome: Incidence of Acute Respiratory Distress Syndrome (ARDS)
Description: Berlin definition of mild ARDS will determine incidence and will be further stratified into Moderate and Severe
Time Frame: Enrollment through 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 100 | 93
Participants | 6 | 3

7. Secondary Outcome: Incidence of Thromboembolic Events
Description: Incidence of pulmonary embolism, venous thrombosis, or arterial thrombosis
Time Frame: Enrollment through 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 100 | 93
Participants | 10 | 10

8. Secondary Outcome: 30-day Mortality
Description: mortality within 30 days
Time Frame: Enrollment through 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
Number analyzed (Participants) | 91 | 82
Participants | 12 | 13

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cold-stored Platelet (CSP) | Standard Care
All-Cause Mortality (participants affected / at risk) | 12/102 | 13/98
Serious Adverse Events (participants affected / at risk) | 9/102 | 4/98
Other Adverse Events (participants affected / at risk) | 0/102 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cold-stored Platelet (CSP) (N=102) | Standard Care (N=98)
Thromboembolic events (Vascular disorders) | 6 (6) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Transfusion Associated Cardiac Overload (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT04667468/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT04667468/ICF_000.pdf